CLINICAL TRIAL: NCT01639560
Title: Varenicline for Light Smokers
Acronym: ChanLight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jon Ebbert, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-005652; WS2293926 (Other Grant/Funding Number: Pfizer Inc)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Smoking
Keywords: smoking; tobacco dependence; nicotine dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): 1 mg of varenicline twice per day for 12 weeks.
  Interventions: Drug: Varenicline
- placebo (Placebo Comparator): 1 placebo tablet twice a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 1 mg of varenicline twice per day for 12 weeks and brief behavioral counseling
  Other Names: chantix
  Arms: Varenicline
Drug: Placebo — 1 placebo tablet twice per day for 12 weeks and brief behavioral counseling
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if varenicline is effective in treating tobacco dependence in adults who smoke 5-10 cigarettes per day.

DETAILED DESCRIPTION:
Nearly 50% of U.S. cigarette smokers smoke ≤ 10 cigarettes per day (CPD) and are considered "light smokers." Most light smokers will either maintain a chronic light smoking habit or increase their level of smoking during their lifetime. Importantly, light smokers are at risk for adverse health consequences and increased all-cause mortality. While multiple factors such as reinforcement behavior, diminished autonomy, economic constraints and tobacco control policies influence light smoking, nicotine dependence appears particularly important in 5 to 10 CPD smokers. Despite the high prevalence of light smoking and its increased healthcare burden, few studies have evaluated the efficacy of pharmacotherapy for this group of smokers. Varenicline, which targets symptoms of nicotine dependence, has been shown to increase smoking abstinence rates in moderate to heavy smokers (≥ 10 cigarettes per day). However, varenicline has not been evaluated in subjects who smoke < 10 CPD. In the current proposal we will investigate the efficacy of varenicline for smoking cessation in 5 to 10 CPD light smokers who wish to quit. This study will be conducted as a double-blind, placebo-controlled, randomized clinical trial at the Mayo Clinic, enrolling 224 eligible participants who smoke 5 to 10 CPD. Participants will receive behavior therapy and either varenicline or placebo for 12 weeks with follow up through 26 weeks. We will determine if varenicline increases smoking abstinence in light smokers at end-of-treatment and 26 weeks as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥ 18 years of age;
2. smokes 5 to 10 CPD for at least 6 months;
3. express interest in quitting smoking;
4. indicate ability to complete all study visits; and
5. provide written informed consent to participate in the study.
6. Subject is a female subject of non-childbearing potential or a female subject of childbearing potential - who is using contraceptives and has a negative pregnancy test result;
7. Subject is in good health as determined by the investigator;
8. Subject has the ability to participate fully in all aspects of the study and keep scheduled appointments.

Exclusion Criteria:

1. An active medical condition such as unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia;
2. History of renal failure;
3. Cancer [excluding non-melanoma skin cancer] not in remission;
4. Psychosis or bipolar disorder;
5. Current unstable or untreated moderate or severe depression as assessed by the CES-D;
6. have, as defined by the C-SSRS (Columbia-Suicide Severity Rating Scale), current non-specific suicidal thoughts, or have a lifetime history of a suicidal attempt (defined as "potentially self-injurious act committed with at least some wish to die, as a result of act.");
7. Substance dependence other than nicotine, defined as:

   a. Patient has a recent history (past month) of heavy alcohol consumption as defined by NIAAA: i. Men: More than 4 drinks on any day or 14 per week ii. Women: More than 3 drinks on any day or 7 per week. b. Use of cocaine, heroin, club drugs (i.e., MDMA/"ecstasy"), methamphetamine, or hallucinogens (e.g., LSD) at any time during the past month.

   c. Use of marijuana on a weekly basis for the past month
8. An allergy to varenicline;
9. Current use of a behavioral or pharmacologic tobacco dependence treatment and unwilling or unable to discontinue use;
10. Another member of their household already participating in this study; and
11. Current treatment with another investigational drug (within 30 days of study entry).
12. Has an unstable medical condition;
13. Subject has untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100;
14. Women of child-bearing potential, or who are pregnant, lactating or likely to become pregnant during the trial and are unwilling to use an acceptable form of contraception during the medication phase will also be excluded. All female subjects of childbearing potential must have a negative pregnancy test and must agree to use approved contraception during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O. Ebbert, MD, Principal Investigator — Mayo Clinic; Ivana T. Croghan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ebbert JO, Croghan IT, Hurt RT, Schroeder DR, Hays JT. Varenicline for Smoking Cessation in Light Smokers. Nicotine Tob Res. 2016 Oct;18(10):2031-5. doi: 10.1093/ntr/ntw123. Epub 2016 Apr 26. PMID 27117285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 45 | 48
End of Treatment | 28 | 20
Completed | 26 | 19
Not Completed | 19 | 29
Not completed — Withdrawal by Subject | 9 | 14
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 9 | 11
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 45 | 48 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 92
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11.7) | 37.2 (11.3) | 37.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 34 | 56
  Male | 23 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 45 | 45 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 0 | 4
  White | 36 | 48 | 84
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 48 | 93
Baseline smoking rate (cigarettes per day) [Mean (Standard Deviation); unit: cigarettes per day] | 7.9 (1.5) | 7.5 (1.5) | 7.7 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Smoking Outcome at 12 Weeks (End of Treatment)
Description: To determine the efficacy of 12 weeks of varenicline therapy in achieving increased smoking abstinence rates in light smokers. Point prevalence is defined as no smoking in the past 7 days.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 45 | 48
participants | 24 | 7
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.7, 95% CI 2-sided [2.5 to 18.1]

2. Primary Outcome: Prolonged Smoking Outcome at 12 Weeks (End of Treatment)
Description: To determine the efficacy of 12 weeks of varenicline therapy in achieving increased smoking abstinence rates in light smokers. Prolonged abstinence is defined as no smoking since 2 weeks after the target quit date.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 45 | 48
participants | 18 | 4
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 7.33, 95% CI 2-sided [2.2 to 24.0]

3. Secondary Outcome: Point Prevalence Smoking Outcome at 24 Weeks (End of Study)
Description: To determine the efficacy of 12 weeks of varenicline therapy in achieving increased smoking abstinence rates at 6 months in light smokers. Point prevalence is defined as no smoking in the past 7 days.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 45 | 48
participants | 18 | 10
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.047, Regression, Logistic; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.0 to 6.3]

4. Secondary Outcome: Prolonged Smoking Outcome at 24 Weeks (End of Study)
Description: To determine the efficacy of 12 weeks of varenicline therapy in achieving increased smoking abstinence rates at 6 months in light smokers. Prolonged abstinence is defined as no smoking since 2 weeks after the target quit date.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 45 | 48
participants | 14 | 4
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 5.0, 95% CI 2-sided [1.5 to 16.5]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected for the entire 6 months of study. Non-serious adverse events were collected for the 3 month-treatment phase.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/48
Other Adverse Events (participants affected / at risk) | 18/45 | 4/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=45) | Placebo (N=48)
Nausea (Gastrointestinal disorders) | 10 (10) | 0 (0)
sleep disturbance (General disorders) | 7 (7) | 1 (1)
Mood Disturbance (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Gastro-esophageal reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of appetite (General disorders) | 1 (1) | 0 (0)
Taste Disturbance (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No